CLINICAL TRIAL: NCT07151651
Title: Endoscopic Lumbar Discectomy: A Comparative Study Between Uniportal and Biportal Endocopic Techniques on Clinical and Surgical Outcomes
Brief Title: A Comparison Between Biportal and Uniportal Endoscopic Lumbar Discectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ibraheem Amin, Assistant lecturer at neurosurgery department sohag University, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sohag-Med-25-8---4MD
Record Dates: First submitted 2025-08-19; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Lumbar Disc Herniation
Keywords: Lumar discectomy; Endoscopy; Uniportal; Biportal
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Intervention Model Description: A prospective study will be conducted at Sohag and Cairo University Hospitals on 60 patients diagnosed with lumbar disc herniation, undergoing endoscopic lumbar discectomy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Patients with lumbar disc prolapse (Active Comparator): 1. Patients aged 18-70 years.
  2. single-level lumbar disc herniation (L3-L4, L4-L5, or L5-S1) confirmed by MRI.
  3. Persistent symptoms not responding to conservative management (≥6 weeks).
  Interventions: Procedure: Endoscopic lumbar discectomy

INTERVENTIONS:
Procedure: Endoscopic lumbar discectomy — Uniportal and boportal endoscopic lumbar discectomy (transforaminal or interlaminar)

SUMMARY:
This study aims to provide a detailed comparison between different methods of lumbar discectomy by the use of different types of spine endoscopy to evaluate the benefits and drawbacks of each type

DETAILED DESCRIPTION:
The aim of this study is to compare between uniportal and biportal endoscopic techniques in patients with lumbar disc herniation in terms of efficacy, safety, and learning curve of endoscopic spine surgery .The research will focus on clinical outcomes, functional recovery, complication rates, patient satisfaction and surgical proficiency in different endoscopic spine surgery techniques, including uniportal and biportal approaches assessing their relative advantages and limitations.

ELIGIBILITY:
Inclusion Criteria:

* All patients should fulfill the following criteria

  1. Patients aged 18-70 years.
  2. single-level lumbar disc herniation (L3-L4, L4-L5, or L5-S1) confirmed by MRI.
  3. Persistent symptoms not responding to conservative management (≥6 weeks).

Exclusion Criteria:

* All patients should not have any of the following criteria

  1. Multilevel disc herniation.
  2. Previous lumbar spine surgery, trauma or injection.
  3. Severe spinal stenosis.
  4. Severe osteoporosis, infection, or malignancy or autoimmune disease affecting the spine.
  5. Uncontrolled medical comorbidities contraindicating surgery.
  6. Instability: spondylolisthesis>grade 1
  7. Marked obesity.(BMI >35-40 kg/m2 )

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measures After endoscopic lumbar discectomy Pain relief | 12 weeks up to 2 years
  1-Pain Relief: Visual Analog Scale (VAS for leg and back pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University, Sohag, Sohag Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Data is not collected yet